CLINICAL TRIAL: NCT04081532
Title: The Effectiveness of Laparoscopic Treatment of Isolated Superficial Peritoneal Endometriosis for Managing Chronic Pelvic Pain in Women: a Randomised Controlled Feasibility Trial
Brief Title: The Effectiveness of Laparoscopic Treatment of Superficial Endometriosis for Managing Chronic Pelvic Pain
Acronym: ESPriT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Grampian (Other Government); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AC19062
Record Dates: First submitted 2019-08-15; First posted 2019-09-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: endometriosis; laparoscopy; pelvic pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: General Practitioner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment (Active Comparator)
  Interventions: Procedure: surgical removal of superficial peritoneal endometriosis
- No surgical treatment (No Intervention)

INTERVENTIONS:
Procedure: surgical removal of superficial peritoneal endometriosis — In the active comparator group patients will have endometriosis lesions removed by ablation or excision. Patients randomised to no surgical treatment arm will not have lesions removed and will only be given diagnosis on whether endometriosis was found or not.
  Arms: Surgical treatment

SUMMARY:
Endometriosis is a chronic, incurable condition that affects about 10% of women of reproductive age. It is defined as a growth of cells similar to the womb lining outside of the womb in the pelvis, and is associated with chronic pelvic pain, excessive period pain, pain with sexual intercourse and difficulties in getting pregnant. If the disease is found only on the lining of the pelvis it is known as "superficial peritoneal" and is usually treated during a laparoscopic surgery by cutting out (excision) or burning off (ablation). However, many women do not find improvement in their symptoms after the surgery and can have complications from the procedure. The aim of this study is to determine if removal of the superficial peritoneal endometriosis improves pain symptoms and quality of life, which method of removal (excision or ablation) is more effective or if surgical removal is of no benefit to the patients and can potentially cause harm. The investigators plan to recruit up to 90 women from four NHS hospitals in Scotland over a period of 12 months. Women who are attending gynaecology departments with pelvic pain who have not previously had a diagnosis of endometriosis via laparoscopy will be approached. Patients will be asked to read an information sheet about the trial. Women who consent to the trial will be randomised during the surgery, if superficial endometriosis is found, to either having the endometriosis removed or not. For this pilot, follow up will be at 3 and 6 months (and obtain permission to continue to follow them up at 12 and 24 months should time and finding permit). Patients who do not consent to take part in the trial will be asked if the investigators can collect data on their demographics and reasons on why they did not wish to take part.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopy for the investigation of chronic pelvic pain
* In order to be randomised, isolated superficial peritoneal endometriosis (SPE) must be identified at laparoscopy (macroscopically)
* Able to give informed consent

Exclusion Criteria:

* Previous surgical diagnosis of endometriosis
* Pregnant or are actively trying for pregnancy within the next six months
* Deep endometriosis or ovarian endometrioma on imaging or at laparoscopy
* Peritoneal 'pockets' only noted at laparoscopy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women with suspected SPE undergoing diagnostic laparoscopy that were approached for the study an agreed to randomisation | Screening
  The proportion of screened women who are eligible for the trial determined from the screening logs

SECONDARY OUTCOMES:
Baseline characteristics of eligible women that agree to be randomised and those that decline participation | Screening
  Baseline characteristics including age, social deprivation, ethnicity and duration of pain collected from screened women
Proportion of women having laparoscopy for investigation of chronic pelvic pain that are eligible (i.e. have only SPE) for the trial | visit 2 (day of surgery)
  The proportion of women undergoing diagnostic laparoscopy who go on to be diagnosed with SPE
Effects of treatment and variability in treatment outcomes | visit 2 (day of surgery), 30 days post surgery
  Intraoperative and postoperative complications
Improvement in quality of life | 30 days post surgery, follow up at 3 and 6 months
  Endometriosis Health Profile-30 (EHP-30)
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Rome IV criteria
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Pelvic Pain and Urgency/Frequency Patient (PUF) Symptom Scale
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  PainDetect TM
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Brief Fatigue Inventory (BFI)
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Pain Catastrophising Questionnaire (PCQ)
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Fibromyalgia Scale
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Measure Yourself Medical Outcome Profile 2 (MYMOP 2)
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  Working Productivity and Activity Impairment Questionnaire (WPAIQ)
Improvement in quality of life | day of surgery, follow up at 3 and 6 months
  EuroQol 5 Dimensions 5 Level Questionnaire (EQ-5D-5L)
Effects of treatment and variability in treatment outcomes | 30 days post surgery, follow up at 3 and 6 months
  Number of patients who needed analgesia after laparoscopy recorded during follow up.
Effects of treatment and variability in treatment outcomes | 30 days post surgery, follow up at 3 and 6 months
  Number of patients who needed medical management with ovarian suppression after laparoscopy recorded during follow up.
Effects of treatment and variability in treatment outcomes | Throughout the trial starting from day of surgery until end of followup at 6 months
  Adverse events (as reported by the participants)
To determine the most acceptable methods of recruitment and assessment tools | Questionnaires collected at Baseline (within a week of surgery), 3 and 6 months follow up
  The proportion of completed trial questionnaires
To determine the most acceptable methods of assessment tools | Throughout the trial until end of follow up at 6 months
  Number of patients who remained blinded for 6 months after the surgery recorded by asking patient if they were told their allocation
To determine the most acceptable methods of recruitment, randomisation and assessment tools | 6 months follow up
  Acceptability of the trial completed at 6 months after surgery will be compared between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Horne, Prof, Study Chair — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Whitaker LHR, Doust A, Stephen J, Norrie J, Cooper K, Daniels J, Hummelshoj L, Cox E, Beatty L, Chien P, Madhra M, Vincent K, Horne AW. Laparoscopic treatment of isolated superficial peritoneal endometriosis for managing chronic pelvic pain in women: study protocol for a randomised controlled feasibility trial (ESPriT1). Pilot Feasibility Stud. 2021 Jan 7;7(1):19. doi: 10.1186/s40814-020-00740-9. PMID 33413677